CLINICAL TRIAL: NCT02099799
Title: The Effect of Physical Activity Promotion on Short and Long-term Outcomes in COPD
Acronym: WEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O1150-R
Record Dates: First submitted 2014-03-20; First posted 2014-03-31 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: COPD; Emphysema; Chronic Bronchitis
Keywords: Physical Activity; COPD Self-Management; Internet; 6-Minute Walk Test; COPD Exacerbation; Health-related Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistant who assesses outcomes is blinded to randomization group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pedometer and Internet Website (Active Comparator): Pedometer and website with feedback, goal setting, educational and motivational content, and community forum.
  Interventions: Behavioral: Pedometer and Website
- Usual Care (No Intervention): Verbal instructions and written materials about exercise.

INTERVENTIONS:
Behavioral: Pedometer and Website — Pedometer and website with feedback, goal setting, educational and motivational content, and community forum.
  Arms: Pedometer and Internet Website

SUMMARY:
COPD currently afflicts 24 million US residents; the prevalence of COPD is high among Veterans. Persons with COPD have significant functional disability as a result of the disease. This project will determine whether a novel Internet-mediated walking program coupled with a pedometer can improve exercise capacity, improve health-related quality of life, and decrease the risk of acute exacerbations in persons with COPD. If successful, based on estimates that 33 to 64% of COPD patients are Internet users, the proposed exercise intervention could help over 8 million persons. The Veterans Health Administration (VHA) has a strong commitment to providing care to persons with COPD and supporting research directed at COPD-related disability. The 2012-2016 Strategic Plan of the VHA Office of Research and Development includes research in COPD rehabilitation. The proposed research addresses Rehabilitation R&D Service's current priority area of improving disabled Veterans' health-related quality of life by reducing disease burden and maximizing functional recovery.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major cause of global morbidity and is projected to become the third leading cause of death in the world by 2020. In Veterans, the prevalence is high; in VISN1 in FY 2012, 9% of outpatient Veterans had the ICD-9 diagnosis of COPD. In COPD, shortness of breath leads to physical inactivity and significant disability. A growing body of knowledge has identified physical activity and exercise as a modifiable factor that may impact COPD-related morbidity and mortality. Epidemiological and cross-sectional studies have shown that persons with COPD who are more physically active have better functional status and are less likely to be hospitalized and to die. A higher daily step count, when directly measured, is associated with lower risk of acute exacerbations (AEs) and mortality in COPD, independent of lung function. Despite the potential benefits, there have been few interventions to increase walking in persons with COPD. Although supervised pulmonary rehabilitation programs improve exercise capacity, they are not accessible to all who could benefit from them and have low adherence rates.

Novel interventions that incorporate strategies for behavioral change and that are accessible, individualized, and sustained are needed to promote physical activity in persons limited by COPD. Funded by a RR&D CDA-2 Dr. Moy and her team have developed and piloted a novel exercise intervention that combines a website with a pedometer to promote walking in persons with COPD. The program, Every Step Counts (ESC) for Lung Health, accurately monitors walking, provides iterative feedback and individualized goal-setting, and delivers education and motivation.

This study proposes a 2-arm randomized, controlled trial to study the efficacy of ESC to improve exercise capacity in persons with COPD, compared to usual care (verbal and written instructions to exercise).

Primary Aim: Determine the efficacy of the ESC intervention to increase 6-minute walk test (6MWT) distance.

Secondary Aims: Estimate the effect of the ESC intervention on (a) health-related quality of life (HRQL), as measured by the St. George's Respiratory Questionnaire (SGRQ), (b) dyspnea, (c) inflammatory biomarkers C-reactive protein (CRP) and interleukin-6 (IL-6), (d) risk for AEs and COPD-related hospitalizations, and (e) engagement in physical activity as measured by daily step count.

185 subjects will be enrolled for a total of 12 months, with the interventional phase being 6 months followed by an observational phase of 6 months. Subjects will be randomized (1:1 ratio) to one of 2 arms: (1) verbal and written instructions to exercise at home (usual care) or (2) usual care plus pedometer and Internet-mediated walking program. Subjects will perform 6MWTs, complete questionnaires, and have blood drawn at clinic visits at baseline, 3, 6, and 12 months. Telephone contact will occur at 9 months. AE history and daily step count will be assessed at each contact. Analysis of variance will compare 6MWT distance in the intervention and usual care group at 6 months. Multivariate regression models will assess 6MWT distance as a function of treatment group, adjusting for baseline 6MWT distance, study site, season of enrollment, and any unbalanced baseline characteristics.

This study hypothesizes that persons randomized to ESC will have greater 6MWT distance at 6 months, compared to persons in the usual care group. It also hypothesize that persons randomized to ESC will have greater improvements in HRQL, dyspnea, daily step counts, and greater decreases in levels of inflammatory biomarker and risk for AEs and COPD-related hospitalizations, compared to control.

The proposed intervention has the potential to (1) bring an exercise program to the vast majority of persons with COPD who cannot go to a hospital-based pulmonary rehabilitation program, (2) improve the effectiveness of current rehabilitation programs by sustaining long-term exercise, and (3) become an effective and integral part of COPD self-management programs. Ultimately, the intervention could decrease risk of hospitalizations, AEs, and COPD-related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, greater than or equal to 40 years of age
* Clinical diagnosis of COPD defined as either a ratio of FEV1 to forced vital capacity < 0.70 or chest CT evidence of emphysema. CT obtained as part of routine clinical care, independent of research study.
* Medical clearance from healthcare provider to participate in an exercise program
* Have an active email account and can check email at least weekly
* Have access to a computer with Internet connection or willing to come to VABoston or Birmingham VA Medical Center to use study computers
* Pedometer with >90% accuracy compared to manual counts on short clinic walk
* Competent to provide informed consent
* Willingness to make return visits and be available by telephone for duration of study

Exclusion Criteria:

* COPD exacerbation in the previous 1 month
* Unable to ambulate with or without assistance
* Clinical signs of unstable cardiovascular disease or congestive heart failure
* Hypoxemia during 6MWT, i.e. oxygen saturation <85% using supplemental oxygen
* Unable to complete questionnaires
* Unable to collect at least 5 of 7 days of baseline step counts
* Participation in a pulmonary rehabilitation program at time of screening or within the previous 3 months
* Participation in another exercise-related research study at time of screening
* Plans to participate in an exercise-related research study in the next 6 months
* Plans to enroll in a supervised exercise program, such as pulmonary rehabilitation, in the next 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn L. Moy, MD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (2):
- United States (2):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moy ML, Matthess K, Stolzmann K, Reilly J, Garshick E. Free-living physical activity in COPD: assessment with accelerometer and activity checklist. J Rehabil Res Dev. 2009;46(2):277-86. doi: 10.1682/jrrd.2008.07.0083. PMID 19533541
- [Background] Moy ML, Janney AW, Nguyen HQ, Matthess KR, Cohen M, Garshick E, Richardson CR. Use of pedometer and Internet-mediated walking program in patients with chronic obstructive pulmonary disease. J Rehabil Res Dev. 2010;47(5):485-96. doi: 10.1682/jrrd.2009.07.0091. PMID 20803392
- [Background] Moy ML, Teylan M, Danilack VA, Gagnon DR, Garshick E. An index of daily step count and systemic inflammation predicts clinical outcomes in chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2014 Feb;11(2):149-57. doi: 10.1513/AnnalsATS.201307-243OC. PMID 24308588
- [Background] Danilack VA, Weston NA, Richardson CR, Mori DL, Moy ML. Reasons persons with COPD do not walk and relationship with daily step count. COPD. 2014 Jun;11(3):290-9. doi: 10.3109/15412555.2013.841670. Epub 2013 Oct 23. PMID 24152213
- [Background] Moy ML, Teylan M, Weston NA, Gagnon DR, Danilack VA, Garshick E. Daily step count is associated with plasma C-reactive protein and IL-6 in a US cohort with COPD. Chest. 2014 Mar 1;145(3):542-550. doi: 10.1378/chest.13-1052. PMID 24091482
- [Background] Moy ML, Teylan M, Weston NA, Gagnon DR, Garshick E. Daily step count predicts acute exacerbations in a US cohort with COPD. PLoS One. 2013 Apr 4;8(4):e60400. doi: 10.1371/journal.pone.0060400. Print 2013. PMID 23593211
- [Background] Moy ML, Danilack VA, Weston NA, Garshick E. Daily step counts in a US cohort with COPD. Respir Med. 2012 Jul;106(7):962-9. doi: 10.1016/j.rmed.2012.03.016. Epub 2012 Apr 20. PMID 22521225
- [Background] Moy ML, Garshick E, Matthess KR, Lew R, Reilly JJ. Accuracy of uniaxial accelerometer in chronic obstructive pulmonary disease. J Rehabil Res Dev. 2008;45(4):611-7. doi: 10.1682/jrrd.2007.09.0147. PMID 18712646
- [Background] Moy ML, Collins RJ, Martinez CH, Kadri R, Roman P, Holleman RG, Kim HM, Nguyen HQ, Cohen MD, Goodrich DE, Giardino ND, Richardson CR. An Internet-Mediated Pedometer-Based Program Improves Health-Related Quality-of-Life Domains and Daily Step Counts in COPD: A Randomized Controlled Trial. Chest. 2015 Jul;148(1):128-137. doi: 10.1378/chest.14-1466. PMID 25811395
- [Derived] Berube MN, Robinson SA, Wan ES, Mongiardo MA, Finer EB, Moy ML. Physical Activity and Systemic Biomarkers in Persons With COPD: Insights from a Web-Based Pedometer-Mediated Intervention. Chronic Obstr Pulm Dis. 2024 Jul 25;11(4):369-381. doi: 10.15326/jcopdf.2023.0472. PMID 38809105
- [Derived] Wan ES, Polak M, Goldstein RL, Lazzari AA, Kantorowski A, Garshick E, Moy ML. Physical Activity, Exercise Capacity, and Body Composition in U.S. Veterans with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2022 Oct;19(10):1669-1676. doi: 10.1513/AnnalsATS.202111-1221OC. PMID 35536690
- [Derived] Cruz Rivera PN, Goldstein RL, Polak M, Lazzari AA, Moy ML, Wan ES. Performance of bioelectrical impedance analysis compared to dual X-ray absorptiometry (DXA) in Veterans with COPD. Sci Rep. 2022 Feb 4;12(1):1946. doi: 10.1038/s41598-022-05887-4. PMID 35121763

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from Nov 2015-Nov 2019 at two US sites. VABoston (BOS) and VABirmingham (BIR).
  204 consented (143 BOS and 61 BIR); 51 not randomized (38 ineligible and 13 withdrew); 153 randomized (108 BOS and 45 BIR); 75 allocated to Pedometer and Internet Website Arm (54 BOS and 21 BIR); 15 Lost to follow-up at 6 months (8 BOS and 7 BIR); 74 included in the analyses.
Pre-assignment Details: 51 not randomized (38 ineligible and 13 withdrew)
Period: Overall Study
Arm/Group | Pedometer and Internet Website | Usual Care
Started | 75 | 78
Completed | 60 | 54
Not Completed | 15 | 24

BASELINE CHARACTERISTICS:
Groups:
- Pedometer and Internet Website: Pedometer and Website: Pedometer and website with feedback, goal setting, educational and motivational content, and community forum.
  Participants were recruited from May 2015- February 2019 at two US sites. VABoston (BOS) and VABirmingham (BIR).
  204 consented (143 BOS and 61 BIR) 51 not randomized (38 ineligible and 13 withdrew) 153 randomized (108 BOS and 45 BIR) 75 allocated to Pedometer and Internet Website Arm (54 BOS and 21 BIR) 15 Lost to follow-up at 6 months (8 BOS and 7 BIR) 74 included in the analyses
- Usual Care: Verbal instructions and written materials about exercise. Participants were recruited from May 2015- February 2019 at two US sites. VABoston (BOS) and VABirmingham (BIR).
  204 consented (143 BOS and 61 BIR) 51 not randomized (38 ineligible and 13 withdrew) 153 randomized (108 BOS and 45 BIR) 78 allocated to Pedometer and Internet Website Arm (54 BOS and 24 BIR) 24 Lost to follow-up at 6 months (13 BOS and 11 BIR) 78 included in the analyses
- Total: Total of all reporting groups
Arm/Group | Pedometer and Internet Website | Usual Care | Total
Number analyzed (Participants) | 75 | 78 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (7.2) | 70.4 (7.3) | 69.3 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 70 | 72 | 142
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 69 | 69 | 138
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
6-Minute Walk Test Distance [Mean (Standard Deviation); unit: meters] | 360.8 (92.0) | 357.2 (103.5) | 359 (97.7)
FEV1 percent predicted [Mean (Standard Deviation); unit: percent] | 60.6 (23.1) | 61.5 (19.8) | 61.1 (21.4)
Daily Step Count [Mean (Standard Deviation); unit: steps per day] | 3242 (2177) | 3320 (2278) | 3281 (2222)

OUTCOME MEASURES:

1. Primary Outcome: 6-Minute Walk Test Distance
Description: In-clinic test that measures exercise capacity. Change in 6MWT distance at 6 months compared to baseline.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: meters
Arm/Group | Pedometer and Internet Website | Usual Care
Number analyzed (Participants) | 75 | 78
meters | 25 (10) | 37 (10)
Statistical Analysis 1: Comparison: Pedometer and Internet Website vs Usual Care; Test type: Superiority; p = 0.189, Mixed Models Analysis; Mean Difference (Final Values) = -12

2. Secondary Outcome: Health-related Quality of Life
Description: Questionnaires that assess quality of life. St. George's Respiratory Questionnaire Total Score Scores range 0-100 Higher score reflects worse HRQL. Change at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pedometer and Internet Website | Usual Care
Number analyzed (Participants) | 75 | 78
score on a scale | -13.0 (3.6) | -15.1 (3.2)
Statistical Analysis 1: Comparison: Pedometer and Internet Website vs Usual Care; Test type: Superiority; p = 0.572, Mixed Models Analysis; Mean Difference (Final Values) = 2.1

3. Secondary Outcome: Dyspnea
Description: Assessed by questionnaire that measure breathlessness and shortness of breath. mMRC dyspnea score Scores range 0-4. Higher values reflect more shortness of breath.
  Change at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pedometer and Internet Website | Usual Care
Number analyzed (Participants) | 75 | 78
score on a scale | -0.1 (0.2) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Pedometer and Internet Website vs Usual Care; Test type: Superiority; p = 0.799, Mixed Models Analysis; Mean Difference (Final Values) = -0.1

4. Secondary Outcome: Engagement in Physical Activity
Description: Assessed by daily step counts on pedometer.
  Change at 6 months compared to baseline.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: steps per day
Arm/Group | Pedometer and Internet Website | Usual Care
Number analyzed (Participants) | 75 | 78
steps per day | 673 (392) | -639 (415)
Statistical Analysis 1: Comparison: Pedometer and Internet Website vs Usual Care; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 1312

5. Secondary Outcome: Inflammatory Biomarker Number 1
Description: RAGE-receptor of advanced glycation end-products
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pedometer and Internet Website | Usual Care
Number analyzed (Participants) | 49 | 39
pg/mL | 95.0 (319) | 22.0 (243)
Statistical Analysis 1: Comparison: Pedometer and Internet Website; Test type: Superiority; p = 0.2265, t-test, 2 sided

6. Other Pre Specified Outcome: Inflammatory Biomarker Number 2
Description: Inflammatory protein biomarker NT-proBNP (beta natriuretic peptide)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pedometer and Internet Website | Usual Care
Number analyzed (Participants) | 49 | 39
pg/mL | 57.1 (498) | 69.2 (314)
Statistical Analysis 1: Comparison: Pedometer and Internet Website vs Usual Care; Test type: Superiority; p = 0.8897, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Description: Significant, pulmonary, and musculoskeletal adverse events were tracked during the study. Significant adverse events were defined as deaths and/or hospitalizations. Pulmonary adverse events were self-reported at 3 and 6 months and included diagnoses of pneumonia and/or acute exacerbation of COPD. Musculoskeletal events were self-reported as chest, leg, foot and/or back pain or discomfort. Serious adverse events were defined as deaths and/or hospitalizations.
Arm/Group | Pedometer and Internet Website | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/75 | 1/78
Serious Adverse Events (participants affected / at risk) | 24/75 | 25/78
Other Adverse Events (participants affected / at risk) | 36/75 | 25/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pedometer and Internet Website (N=75) | Usual Care (N=78)
Hospitalizations (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 24 (24) — Mainly for COPD acute exacerbations
Death (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — One death from leukemia. The cause of the other death is unknown.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pedometer and Internet Website (N=75) | Usual Care (N=78)
Musculoskeletal adverse event (Musculoskeletal and connective tissue disorders) | 36 (36) | 25 (25)

LIMITATIONS AND CAVEATS:
Strengths include the randomized study design, dual-site approach, and 6-month time frame. While the study expanded our past work with a more socioeconomically diverse sample, our cohort was self-selected and majority male, limiting generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT02099799/Prot_SAP_000.pdf